CLINICAL TRIAL: NCT01633229
Title: A Phase I Study of Bone Marrow Stromal Cell Infusions to Treat Acute Graft Versus Host Disease, Marrow Failure and Tissue Injury After Allogeneic Stem Cell Transplantation
Brief Title: Bone Marrow Stromal Cell Infusions for Stem Cell Transplant Complications
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120010; 12-H-0010
Record Dates: First submitted 2012-06-30; First posted 2012-07-04 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2018-03-08

CONDITIONS: Graft-Versus-Host Disease
Keywords: Immune Suppression; BMSC; GVHD; Marrow Failure; Regimen Related Toxicity; Graft-Versus-Host Disease
MeSH Terms: conditions — Graft vs Host Disease

INTERVENTIONS:
Procedure: Bone Marrow Stromal Cell Infusion

SUMMARY:
Background:

* Bone marrow stromal cells (BMSC) from bone marrow biopsies can be used to treat disorders that cause inflammation and immune system diseases. BMSC have been used to treat graft versus host disease (GVHD), a complication that can develop after stem cell transplants. BMSC have also been used to treat other post-transplant complications, like marrow failure or tissue injury.
* The National Institutes of Health (NIH) has developed a procedure for collecting and preserving BMSC from volunteer donors. These donors have passed tests to ensure that their cells are healthy enough to be used for treatment. Researchers want to use the collected cells to treat people with GVHD, marrow failure, or tissue injury following stem cell transplants.

Objectives:

- To test the safety and effectiveness of NIH-collected BMSC to treat complications from stem cell transplants.

Eligibility:

* Individuals between 18 and 75 years of age who have complications from stem cell transplants.
* Complications are acute GVHD, poor bone marrow function, or tissue or organ damage.

Design:

* Participants will be screened with a physical exam and medical history. They will also have imaging studies and blood tests.
* Participants will provide blood, skin, and bone marrow samples before the BMSC treatment. Additional samples, including tissue samples, will be collected after the start of treatment.
* Participants will have up to three BMSC infusions. There will be a week between each infusion. Participants will be monitored closely during each infusion. Any side effects will be treated.
* Treatment will be monitored with frequent blood tests and physical exams.
* After the end of the infusions, participants will have regular followup visits for up to 2 years.

DETAILED DESCRIPTION:
Bone marrow stromal cells (BMSC) derived from bone marrow aspiration/biopsy have important anti-inflammatory and immunosuppressive properties that make them suitable candidates for cellular therapy of inflammatory and degenerative disorders. BMSC suppress lymphocyte immune responsiveness and can hone in to sites of inflammation and promote healing. BMSC were first used in man to successfully treat refractory acute graft versus host disease (aGVHD). A recent multicenter study treating refractory aGVHD reported a 66% response rate and a sustained survival in responding patients. BMSC are currently being evaluated in acute GVHD in several ongoing studies worldwide. BMSC have also been used to treat post-transplant conditions not directly due to GVHD. Responses have been reported in hemorrhagic cystitis, and pneumoperitoneum. BMSC are also under evaluation in the treatment of inflammatory and autoimmune disorders.

The Cell Processing Section of the Department of Transfusion Medicine at the Clinical Center NIH has developed a procedure for collecting, expanding and cryopreserving clinical grade BMSC under an FDA Drug Master File (DMF). Marrow will be aspirated from volunteer donors participating on protocol 10-CC-0053 who have passed the standard screening for blood and marrow donors and BMSC will be expanded in vitro. Since it is not necessary to HLA-match BMSC donors with their recipient for this study, a BMSC repository will be used as the source of BMSC for this study.

This will be the first trial of the safety of the NIH BMSC cellular product in stem cell transplant recipients. In this phase I study, open to adult NIH allogeneic stem cell transplantation (SCT) recipients, we will evaluate the safety of a fixed dose of BMSC infusions (target dose of 2 x 106 BMSCs /kg (+/- 10%)) in patients with acute GVHD, marrow failure or tissue injury following allogeneic SCT. Up to three BMSC infusions will be given every 7 3 days apart. Safety will be monitored continuously with a stopping rule for toxicity based on the treatment-related serious adverse event rate. Organ-specific clinical responses will be measured. Where possible we will also attempt to identify transfused BMSC in sites of damage in biopsy material. It is planned to accrue up to 10 subjects over a 6-month period.

ELIGIBILITY:
* INCLUSION CRITERIA:

5.1.1 History of allogeneic SCT

Any subject who has received an allogeneic SCT at NIH is eligible if they have one or more of the following conditions. Subjects may continue to receive standard treatments for their condition but may not be entered onto a new investigational protocol to treat the condition during the period of evaluation of BMSC infusions.

5.1.1.1 Acute GVHD

Biopsy confirmed within 14 days of investigational intervention (unless not possible to perform because of anatomical location or clinical contraindication) acute GVHD affecting gut and/or liver and/or skin, defined as steroid refractory: failure to respond to greater than or equal to 2mg/kg methylprednisolone (or equivalent) after 7 days OR steroid dependent: requiring methylprednisolone (or equivalent) greater than or equal to 1mg/kg for greater than or equal to 7days for control of GVHD. GVHD affecting the skin alone is rarely lethal and is excluded. Acute GVHD is defined using the NIH consensus definition inclusive of Classic acute (< 100 days after transplant or DLI, presence of acute GVHD features, absence of chronic GVHD features) AND Persistent/recurrent/late onset acute (> 100 days after transplant or DLI, presence of acute GVHD features, absence of chronic GVHD features).

5.1.1.2 Marrow Failure

Poor graft function in the presence of >95% donor myeloid chimerism: defined as platelet or red cell transfusion dependent OR absolute neutrophil count persisting <500/ (Micro)l for 14 days without other reversible or treatable causes.

5.1.1.3 Pulmonary injury

Lung injury from: Diffuse alveolar hemorrhage (DAH), Cryptogenic Organizing Pneumonia (COP), Bronchiolitis Obliterans Syndrome (BOS), idiopathic interstitial pneumonia (IP), Adult respiratory distress syndrome (ARDS) diagnosed by exclusion of active infection. Also worsening pneumomediastinum or pneumothorax persisting after 7 days; at risk for causing hemodynamic changes in association with any of these diagnoses.

5.1.1.4 Hepatic injury

Clinically diagnosed sinusoidal obstruction syndrome (SOS), previously known as veno-occlusive disease (VOD), with bilirubin > 2 times ULN or transaminases >3 times ULN and rising.

5.1.1.5 Hemorrhagic cystitis (HC)

HC requiring continuous bladder irrigation OR requiring red cell or platelet transfusions at least intermittently for the past 7 days OR HC unresponsive to antivirals after 10 days.

5.1.1.6 Gastrointestinal tract

Pneumoperitoneum, bowel perforation not susceptible to corrective surgery OR blood transfusion requirement > 1 unit per day for 7 days.

5.1.2 Age: greater than or equal to 18 years of age and less than or equal to 75 years of age.

5.1.3 Birth Control

Subjects of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are being treated on this study.

5.1.4 Transplant performed at NIH.

EXCLUSION CRITERIA:

5.2.1 Breast feeding or pregnant females (due to unknown risk to fetus or newborn).

5.2.2 Allergic to gentamicin

5.2.3 Weight less than 20 kg (not informative for research sampling)

5.2.4 Patients with significant organ failure at baseline as evidenced by any of the following:

1. <TAB>Symptomatic cardiac failure at rest or with minimal activity or exertion for which intervention is indicated
2. <TAB>Creatinine > 3.0 X ULN
3. <TAB>Decreased oxygen saturation at rest (e.g. pulse oximeter < 88% or PaO2 less than or equal to 55 mmHg)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-11-14; Primary Completion 2013-07-01 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint to this study is to characterize the safety of bone marrow stromal cells (BMSC).

CONTACTS AND LOCATIONS:
Overall Officials: Minocher M Battiwalla, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ogawa M, LaRue AC, Drake CJ. Hematopoietic origin of fibroblasts/myofibroblasts: Its pathophysiologic implications. Blood. 2006 Nov 1;108(9):2893-6. doi: 10.1182/blood-2006-04-016600. Epub 2006 Jul 13. PMID 16840726
- [Background] Bhanu NV, Trice TA, Lee YT, Gantt NM, Oneal P, Schwartz JD, Noel P, Miller JL. A sustained and pancellular reversal of gamma-globin gene silencing in adult human erythroid precursor cells. Blood. 2005 Jan 1;105(1):387-93. doi: 10.1182/blood-2004-04-1599. Epub 2004 Sep 14. PMID 15367428
- [Background] Taylor HS. Endometrial cells derived from donor stem cells in bone marrow transplant recipients. JAMA. 2004 Jul 7;292(1):81-5. doi: 10.1001/jama.292.1.81. PMID 15238594